CLINICAL TRIAL: NCT01084330
Title: A Randomized, Open-label, Multi-center Phase II Study to Compare AUY922 With Docetaxel or Irinotecan in Adult Patients With Advanced Gastric Cancer, Who Have Progressed After One Line of Chemotherapy
Brief Title: Phase II Trial of AUY922 vs. Comparators in Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A2202; 2009-015407-47 (EudraCT Number)
Record Dates: First submitted 2010-03-05; First posted 2010-03-10 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-08

CONDITIONS: Advanced Gastric Cancer; Gastro-esophageal Junction Cancer
Keywords: gastric cancer; metastatic gastric cancer; advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Docetaxel; Irinotecan

ARMS (2):
- AUY922 (Experimental)
  Interventions: Drug: AUY922
- Docetaxel or Irinotecan (Active Comparator)
  Interventions: Drug: Docetaxel; Drug: Irinotecan

INTERVENTIONS:
Drug: AUY922 — 70mg/m2
  Arms: AUY922
Drug: Docetaxel — Docetaxel 75mg/m2
  Arms: Docetaxel or Irinotecan
Drug: Irinotecan — Iriniotecan 350mg/m2
  Arms: Docetaxel or Irinotecan

SUMMARY:
A clinical trial to determine the effectiveness and safety of AUY922 compared to other drugs known to be effective against gastric cancer in second line therapy for patients who have failed one line of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed advanced gastric cancer
* One previous line of chemotherapy
* Progressive disease
* One measurable lesion
* Blood tests within protocol ranges
* (WHO) Performance Status ≤ 1
* Able to sign informed consent

Exclusion Criteria:

* No symptomatic brain metastases
* No coumarin type anticoagulants
* No liver or kidney disease
* No impaired heart function
* No pregnant or lactating women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 21 day cycle: treatment until death, lost to follow up or withdrawal

SECONDARY OUTCOMES:
Estimate of the Overall Survival Treatment Effect to see if there is a difference in treatment effect in patients who receive AUY922 versus patients who receive comparator medications. | 21 day cycle: treatment until death, lost to follow up or withdrawal
Objective Response Rate to see if there is a difference in treatment effect in patients who receive AUY922 versus patients who receive comparator medications. | 21 day cycle: treatment until death, lost to follow up or withdrawal
Evaluate Safety by measuring cardiac safety, recording Adverse Events (AEs) and tracking the tolerability of AUY922 | 21 day cycle: treatment until death, lost to follow up or withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (33):
- United States (7):
  - USC/Kenneth Norris Comprehensive Cancer Center USC/Norris, Los Angeles, California
  - University of California at Los Angeles Dept. of UCLA (4), Los Angeles, California
  - Horizon Oncology Center, Lafayette, Indiana
  - The Sidney Kimmel Cancer Center at Johns Hopkins Hospital Dept. of SKCC @ JHU, Baltimore, Maryland
  - Clinical Research Alliance Dept.ofArenaOncologyAssoc(2), Lake Success, New York
  - Baylor Health Care System/Sammons Cancer Center Baylor Texas Oncology, Dallas, Texas
  - Tyler Cancer Center Dept.ofTylerCancerCtr. (2), Tyler, Texas
- Novartis Investigative Site, Adelaide, South Australia, Australia
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Ulm
- Italy (5):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
- Novartis Investigative Site, Bellinzona, Switzerland
- Taiwan (3):
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Ankara, Turkey (Türkiye)
- United Kingdom (4):
  - Novartis Investigative Site, Surrey, England
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leicester

REFERENCES:
- See also: ESMO Abstract — http://www.embase.com/search/results?subaction=viewrecord&rid=3&page=1&id=L71716851
- See also: Results for CAUY922A2202 can be found on the Novartis Clinical Trial Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8643